CLINICAL TRIAL: NCT02660606
Title: A Qualitative Study to Assess the Content Validity of the Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)
Brief Title: A Qualitative Study to Assess the Content Validity of the Prescription Opioid Misuse and Abuse Questionnaire
Acronym: POMAQ
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: Evidera (Industry)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-3; 3033-3 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Group 1: Opioid abusers
  Interventions: Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)
- Group 2: Abusers of other substances
  Interventions: Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)
- Group 3: Non-opioid abusers
  Interventions: Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)
- Group 4: Non-opioid users
  Interventions: Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)

INTERVENTIONS:
Other: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ)

SUMMARY:
The purpose of this study is to evaluate the patient usability and reliability of the POMAQ survey to evaluate opioid misuse and abuse among adults with chronic moderate to severe pain, including patients who are opioid abusers, non-abusers, as well as non-opioid users

DETAILED DESCRIPTION:
The Food and Drug Administration (FDA) has requested, as part of a post-marketing requirement (PMR) for new drug application (NDA) holders of extended release/long-acting (ER/LA) opioids, to conduct a study to develop and validate a measure of the opioid-related adverse events misuse and abuse among patients with chronic pain prescribed long-term opioid therapy. This measure will be used to assess misuse and abuse in PMR Study 2065-1A and PMR Study 2065-4B.

Currently, no tool exists to meet this need except for the Self-report Misuse, Abuse and Diversion of Prescription (Rx) Opioids questionnaire (SR-MAD) which has undergone several rounds of prior content validation. The SR-MAD has been modified to meet the needs of PMR Studies 2065-1A and 2065-4B, and has been renamed the Prescription Opioid Misuse and Abuse Questionnaire (POMAQ).

This study will seek to further develop and validate the POMAQ using the the Food and Drug Administration (FDA) Guidance for Industry, Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims (FDA 2009) as a reference for conducting qualitative research throughout the process of instrument development to ensure the content validity of a measure and to evaluate the comprehensibility of included questions. This qualitative study to evaluate content validity will be conducted prior to the quantitative study to evaluate construct validity

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients who, based on the Site Investigator's clinical judgment, have chronic moderate to severe pain
3. Willing to provide written informed consent
4. Able to participate in a one-on-one interview
5. Able to read, speak, and understand English and complete all study assessments.

Exclusion Criteria:

1. Cognitive, psychiatric or other impairment based on the Site Investigator's clinical judgment that would interfere with participating in a one-on-one discussion
2. Terminal illness with life expectancy < 6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain recruited from primary care or chronic pain clinics
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2016-01-18 (Actual); Study Completion 2016-01-18 (Actual)

PRIMARY OUTCOMES:
Content validity of POMAQ | Day 1, based upon survey completed at single visit
  Evidence of content validity from patients regarding the interpretation of POMAQ items, ease of completion, the comprehensiveness of instrument, and the appropriateness of the format, response scales, and recall period

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Barsdorf, Ph.D., Study Chair — Pfizer
Locations (1):
- Evidera, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Coyne KS, Schnoll SH, Butler SF, Barsdorf AI, Currie BM, Maziere JY, Pierson RF, Porter LN, Franks CMJ Jr, Farrar JT. Clinical scoring algorithm for the prescription opioid misuse and abuse questionnaire (POMAQ). Curr Med Res Opin. 2022 Jun;38(6):971-980. doi: 10.1080/03007995.2022.2065139. Epub 2022 May 13. PMID 35437075